CLINICAL TRIAL: NCT06608537
Title: A Single-center, Single-arm Phase II Clinical Study Based on FAPI-PET/CT Technology to Predict Pathological Complete Response After Neoadjuvant Chemoradiotherapy for MSS Rectal Cancer
Brief Title: A Clinical Study Based on FAPI-PET/CT Technology to Predict Pathological Complete Response After Neoadjuvant Chemoradiotherapy for MSS Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GIHSYSU-FAPI01
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer
Keywords: FAPI; PET/CT; PD-1; neoadjuvant chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neoadjuvant SCRT followed by Sintilimab plus CAPOX (Experimental): Patients received neoadjuvant treatment consisting of SCRT (a total of 25 Gy in 5 days) followed by sintilimab (3mg/kg intravenous drip on day 1; every 3-week cycle for two cycles) combined with CAPOX (oxaliplatin 130 mg/m2 intravenous infusion over 2 h on day 1, capecitabine 1000 mg/m2 orally twice daily from day 1-14, in every 3-week cycle for two cycles) 1 week later.
  Interventions: Drug: neoadjuvant SCRT followed by Sintilimab plus CAPOX

INTERVENTIONS:
Drug: neoadjuvant SCRT followed by Sintilimab plus CAPOX — Patientsreceived neoadjuvant treatment consisting of SCRT (a total of 25 Gy in 5 days) followed by sintilimab (3mg/kg intravenous drip on day 1; every 3-week cycle for two cycles) combined with CAPOX (oxaliplatin 130 mg/m2 intravenous infusion over 2 h on day 1, capecitabine 1000 mg/m2 orally twice daily from day 1-14, in every 3-week cycle for two cycles) 1 week later.

SUMMARY:
The combination of short course radiotherapy and immunotherapy helps to increase the proportion of pathological complete response after neoadjuvant therapy, providing more patients with the opportunity for organ preservation. However, there is no accurate and unified cCR diagnostic standard in the world. As a new radiotracer, 68Ga-FAPI has been developed and used to target fibroblast activating protein and tumor matrix visualization, which has the advantages of low background uptake, high contrast, few preparation requirements, short post-injection interval, and no influence on blood glucose. Therefore, we will invite you to participate in a clinical study to explore whether the PET parameters of 18F-FDG and 68Ga-FAPI-42 PET/CT can be used to predict pathological responses after neoadjuvant therapy for locally advanced rectal cancer (LARC). The findings will help improve future treatment stratification of LARC, help patients preserve organs and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* With my consent and signed informed consent, willing and able to comply with the planned visit, research treatment, laboratory tests and other test procedures;
* Age 18-75;
* Patients with a pathologically or cytologically confirmed adenocarcinoma of the rectum, all other histological types excluded;
* The distance between the lower margin of the rectal tumor lesion and the anal margin <12cm;
* The physical status score (ECOG) of the Eastern United States Cancer Cooperative Group was 0-1 ;
* T3-4/N+ was evaluated by pelvic enhanced MRI;
* Had not received systemic anti-tumor therapy for colon cancer, including cytotoxic drugs, immune checkpoint inhibitor therapy, molecular targeted therapy, endocrine therapy, etc.;
* Appropriate organ function based on the following laboratory test values obtained during the screening period: White blood cell count ≥3×109/L, neutrophil count ≥1.5×109 /L, platelet count ≥75×109 /L, serum total bilirubin ≤ 1.5× upper limit of normal (UNL), AST (SGOT) or ALT (SGPT) ≤ 2.5×UNL, serum creatinine ≤ 1.5×UNL;
* Female subjects of reproductive age must undergo a negative serum pregnancy test within 3 days prior to the start of the study drug and be willing to use a medically approved highly effective contraceptive method (such as an IUD, contraceptive pill, or condom) during the study period and within 3 months after the last study drug administration; Male subjects whose partners are women of reproductive age should be surgically sterilized or agree to use effective contraception during the study period and for 3 months after the last study dosing;
* Willing and able to comply with research procedures and visit plans.

Exclusion Criteria:

* Whole-body CT, MR, or PET-CT (including at least the chest, whole abdomen, and pelvis) confirms distant metastases (M1);
* Patients with complete intestinal obstruction, active bleeding or perforation requiring emergency surgery;
* The presence of other active malignancies in the past or at the same time (except malignancies that have received curative treatment and have been free of disease for more than 5 years or cancers in situ that can be cured by adequate treatment);
* Thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, and deep vein thrombosis, occurred in the 12 months prior to study entry;
* Myocardial infarction, severe/unstable angina pectoris, NYHA grade 2 or higher cardiac dysfunction, clinically significant supracentricular or ventricular arrhythmia, and symptomatic congestive heart failure in the 12 months prior to enrollment;
* Systemic antibiotic use ≥ 7 days within 4 weeks prior to enrollment, or unexplained fever &gt during screening/prior to first dosing; 38.5°C (as determined by the investigators, fever due to tumor could be included); Had received major operations such as laparotomy, thoracotomy, laparoscopic resection of organs or severe trauma within 2 months before enrollment (the surgical incision should be completely healed before enrollment in this clinical trial);
* Known presence of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) related disease;
* The presence of interstitial lung disease, non-infectious pneumonia or uncontrolled systemic diseases (such as diabetes, hypertension, pulmonary fibrosis and acute pneumonia); Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; Hepatitis C, defined as HCV-RNA above the lower detection limit of analytical methods) or co-infection with hepatitis B and hepatitis C;
* A known or suspected history of allergy to any of the relevant drugs used in the study;
* Pregnant or lactating women; Women of reproductive age who do not use or refuse to use effective non-hormonal contraception (after the last menstrual period < 2 years) or men who are likely to have children;
* The presence of other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of participating in the study or interfere with the study results, as well as patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) prediction accuracy | 3 months
  PCR prediction accuracy was defined as the ratio at which 68Ga-FAPI-42 combined with 18F-FDG PET/CT predicted results in agreement with post-operative pathologic diagnoses.

SECONDARY OUTCOMES:
Prediction accuracy of non-pathological complete response (npCR) | 3 months
  The prediction accuracy of nPCR was defined as the ratio at which 68Ga-FAPI-42 combined with 18F-FDG PET/CT predicted nPCR to be consistent with post-operative pathological diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No